CLINICAL TRIAL: NCT00848484
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Add-On Therapy, 2-Period Cross-Over Clinical Trial to Evaluate the Safety and Efficacy of MK5757 for the Treatment of Cognitive Impairment in Men With Schizophrenia
Brief Title: Treatment of Cognitive Impairment in Men With Schizophrenia (MK5757-005)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 5757-005; 2007_603
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK5757
  Interventions: Drug: MK5757
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK5757 — This is a 2 period, cross-over study. In each of the two treatment periods, each patient will receive the following: Days 1 and 28 MK5757 25 mg capsules three times a day (tid). Days 2 through 14 and Days 29 through 42 MK5757 50 mg capsules tid. Study drug is taken 3 times daily. Each treatment period is 14 days
  Arms: 1
Drug: Comparator: Placebo — This is a 2 period, cross-over study. In each of the two treatment periods, each patient will receive the following: Days 1 and 28 MK5757 one placebo capsules three times a day (tid). Days 2 through 14 and Days 29 through 42 two MK5757 placebo capsules tid. Study drug is taken 3 times daily. Each treatment period is 14 days.
  Arms: 2

SUMMARY:
This study is to evaluate the safety and efficacy of the study drug compared to placebo in the treatment of cognitive impairment in men with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male between 21 and 55 years of age
* Duration of the illness must be longer than 1 year
* Patient's current antipsychotic medication regimen must be stable
* Patient is negative for selected drugs of abuse at Screening
* Must be in a stable living arrangement for at least 3 months prior to screening (not a homeless shelter)

Exclusion Criteria:

* Patient has mental retardation
* Undergone Electroconvulsive Therapy (ECT) treatment within 6 months prior to screening
* Has suicidal attempts or ideation within the last 12 months
* Patient has a history of alcohol/drug dependence within 1 year or alcohol/drug abuse within 12 months of starting the study

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Evaluated: 14-Oct-2008, Last Patient Last Visit: 18-Jun-2009; 6 sites (2 United States, 4 Russia). In total, enrollment lasted approximately 8 months.
Pre-assignment Details: Patients in this cross-over study were randomly assigned to placebo or MK5757 for 2 weeks separated by a 2-week wash-out period. Women were not permitted to enroll into this study because safety, pharmacokinetic or pharmacodynamic properties of MK5757 in women have not been established.
Groups:
- MK5757 / Placebo: Patients were randomly assigned to two weeks of treatment with MK5757 during Treatment Period 1 followed by a 2-week washout followed by administration of placebo during Treatment Period 2.
  Patients received one orally-administered three times a Day[ter in die] (tid) dose on the first day of each treatment period. Patients titrated to two orally-administered tid doses on the second day of each Treatment Period and had the option to down-dose to one tid dose for the remainder of that treatment period.
  Patients who down-dosed during Treatment Period 1 titrated to the target dose of 50 mg tid (or the placebo equivalent) during Treatment Period 2, but were permitted to down-dose if necessary. A 14-day Washout Period separated each 14-day treatment period
- Placebo / MK5757: Patients were randomly assigned to two weeks of treatment with placebo during Treatment Period 1 followed by a 2-week washout followed by administration of MK5757 during Treatment Period 2.
  Patients received one orally-administered three times a Day[ter in die] (tid) dose on the first day of each treatment period. Patients titrated to two orally-administered tid doses on the second day of each Treatment Period and had the option to down-dose to one tid dose for the remainder of that treatment period.
  Patients who down-dosed during Treatment Period 1 titrated to the target dose of 50 mg tid (or the placebo equivalent) during Treatment Period 2, but were permitted to down-dose if necessary. A 14-day Washout Period separated each 14-day treatment period
Period: First Intervention (Treatment Period 1)
Arm/Group | MK5757 / Placebo | Placebo / MK5757
Started | 27 | 27
With Reduced Dose at Treatment Period 1 | 2 | 1
Completed | 25 | 24
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period of Two Weeks
Arm/Group | MK5757 / Placebo | Placebo / MK5757
Started | 25 | 24
Completed | 25 | 21
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3
Period: Second Intervention (Treatment Period 2)
Arm/Group | MK5757 / Placebo | Placebo / MK5757
Started | 25 | 21
With Reduced Dose at Treatment Period 2 | 0 | 0
Completed | 25 | 20
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK5757 / Placebo | Placebo / MK5757 | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.5) | 36.1 (9.1) | 35.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 27 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 24 | 27 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6 | 7 | 13
  Multi-Racial | 1 | 0 | 1
  White | 20 | 20 | 40
Study Region [Number; unit: participants]
  United States | 8 | 7 | 15
  Russia | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Composite Score From the Brief Assessment of Cognition in Schizophrenia (BACS) Battery After 2 Weeks of Treatment
Description: The Brief Assessment of Cognition in Schizophrenia (BACS) was used to evaluate cognitive impairment, as measured by the mean change from baseline after 2 weeks of treatment in the composite score. The BACS composite score was calculated by averaging scores from the BACS subtests, including Verbal Memory, Digit Sequencing, Token Motor, Symbol Coding, Verbal Fluency (Semantic Fluency and Letter Fluency) and Tower of London. The possible minimum and maximum scores for change from baseline at two weeks of treatment for the endpoint are -111.5 and 111.5, respectively.
Time Frame: Baseline and Week 2
Population: Full Analysis Set (FAS): The FAS population was a subset of all randomized patients which included randomized patients who received at least one dose of study treatment and had at least one measurement in any of the two treatment periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Groups:
- MK5757: MK5757 50 mg tid for Treatment Period 1 or Treatment Period 2 (depending on the sequence). Patients who were unable to tolerate 50 mg tid were allowed to titrate down to 25 mg tid and remained on 25 mg tid for the remainder of the treatment period.
- Placebo: Matching placebo 50 mg tid for Treatment Period 1 or Treatment Period 2 (depending on the sequence). Patients who were unable to tolerate 50 mg tid were allowed to titrate down to 25 mg tid and remained on 25 mg tid for the remainder of the treatment period.
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | 0.3 [-1.2 to 1.7] | 1.5 [0.1 to 2.8]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.277, constrained Longitudinal Data Analysis; The repeated measures model included the terms site and sequence * time with a restriction of the same baseline mean across treatment sequences

2. Secondary Outcome: Mean Change From Baseline After 2 Weeks of Treatment in the CogState Composite Score
Description: CogState Schizophrenia Battery was used to evaluate cognitive impairment, as measured by the mean change from baseline after 2 weeks of treatment in the composite score. The composite score was comprised of 4 modules from the CogState Schizophrenia Battery: Identification Task, Detection Task, One Card Learning Task and Groton Maze Learning Task. Composite score was calculated by averaging all available standardized tests scores for the specified tests. The possible minimum and maximum scores for change from baseline at 2 weeks of treatment for the endpoint are -347.5 and 347.5, respectively.
Time Frame: Baseline and week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | 0.3 [-1.7 to 2.4] | -0.5 [-2.5 to 1.5]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.686, constrained Longitudinal Data Analysis — The Benjamini & Hochberg False Discovery Rate (FDR) approach at critical value 0.1 was used to adjust p-Values among five secondary cognition endpoints; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline After 2 Weeks of Treatment in the Executive Functioning Composite Score
Description: The Executive Functioning Composite Score was comprised of the following tests: Groton Maze Learning Task from the CogState Schizophrenia Battery and Tower of London, Semantic Fluency and Letter Fluency tests from the BACS. The composite score was calculated by averaging all of the available standardized tests scores for the specified tests. The possible minimum and maximum scores for change from baseline at two weeks of treatment for the endpoint are -253.4 and 253.4, respectively.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | 0.9 [-0.9 to 2.6] | 1.0 [-0.7 to 2.6]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.933, constrained Longitudinal Data Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Change From Baseline After 2 Weeks of Treatment in the Episodic Memory Composite Score
Description: The Episodic Memory Composite Score was comprised of the following tests: Continuous Paired Associate Learning Task and One Card Learning Task from the CogState Schizophrenia Battery and the Verbal Memory test from the BACS. The composite score was calculated by averaging all of the available standardized tests scores for the specified tests. The possible minimum and maximum scores for change from baseline at two weeks of treatment for the endpoint are -207.06 and 207.06, respectively.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | 0.1 [-1.4 to 1.6] | 0.8 [-0.7 to 2.3]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.686, constrained Longitudinal Data Analysis — The Benjamini & Hochberg False Discovery Rate (FDR) approach at critical value 0.1 was used to adjust p-Values among 5 secondary cognition endpoints; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Change From Baseline After 2 Weeks of Treatment in the Working Memory Composite Score
Description: The Working Memory Composite Score was comprised of the following tests: Two-Back Memory Task from the CogState Schizophrenia Battery and the Digit Sequencing test from the BACS. The composite score was calculated by averaging all of the available standardized tests scores for the specified tests. The possible minimum and maximum scores for change from baseline at two weeks of treatment for the endpoint are -27.06 and 27.06, respectively.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | -1.7 [-3.6 to 0.2] | -0.1 [-1.9 to 1.7]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.686, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Mean Change From Baseline After 2 Weeks of Treatment in the Attention/Processing Speed Composite Score
Description: The Attention/Processing Speed Composite Score was comprised of the following tests: Identification Task and the Detection Task from the CogState Schizophrenia Battery and the Symbol Coding test from the BACS. The composite score was calculated by averaging all of the available standardized tests scores for the specified tests. The possible minimum and maximum scores for change from baseline at two weeks of treatment for the endpoint are -287.15 and 287.15, respectively.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: T-score based on normative data
Arm/Group | MK5757 | Placebo
Number analyzed (Participants) | 42 | 46
T-score based on normative data | -0.2 [-2.1 to 1.6] | -1.3 [-3.1 to 0.4]
Statistical Analysis 1: Comparison: MK5757 vs Placebo; Test type: Superiority or Other; p = 0.686, constrained Longitudinal Data Analysis — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All clinical adverse events within 14 days post dose and all laboratory adverse events post dose are included.
Description: The number of patients listed in the Adverse Event tables is the number of
  patients who received study treatment and had follow-up.
Arm/Group | MK5757 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/52
Other Adverse Events (participants affected / at risk) | 15/48 | 8/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK5757 (N=48) | Placebo (N=52)
Electrocardiogram QT prolonged (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK5757 (N=48) | Placebo (N=52)
Sinus bradycardia (Cardiac disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Electrocardiogram change (Investigations) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 3
Somnolence (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.